CLINICAL TRIAL: NCT01280786
Title: A Phase 1 Dose-Escalation Study of Elesclomol Sodium Administered Intravenously to Subjects With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Study Elesclomol Sodium in Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Synta 4783-14
Record Dates: First submitted 2011-01-14; First posted 2011-01-21 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; leukemia; relapsed or refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elesclomol Sodium (Experimental)
  Interventions: Drug: Elesclomol Sodium

INTERVENTIONS:
Drug: Elesclomol Sodium — Weekly intravenous administration of escalating doses of elesclomol sodium provided response is seen after the first 4 week cycle.

SUMMARY:
This is a phase 1 study to test the safety of escalating doses of elesclomol sodium given to patients with advanced myeloid leukemia.

DETAILED DESCRIPTION:
This aim of this study is to determine the safety and tolerability of elesclomol sodium at escalating doses (ultimately identifying the maximum tolerated dose) when administered to patients with advanced myeloid leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Adults with cytologically confirmed Acute Myeloid Leukemia (AML) that has relapsed after the completion of induction and/or consolidation therapy or has failed to respond to standard induction therapy
* ECOG performance status of 0-2
* Acceptable organ and marrow function during the screening period as defined by the protocol
* Reliable venous access suitable for study drug infusions

Exclusion Criteria:

* Significant cardiovascular disease
* Candidates for hematopoietic stem cell transplant
* Women who are pregnant or breast-feeding
* Prior treatment with chronic immunosuppressants
* Other clinically significant uncontrolled conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-06 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of adverse events based on frequency, causality, and severity as a measure of safety and tolerability. | 1 year
  - Characterize the safety and tolerability of elesclomol sodium administered to subjects with relapsed or refractory acute myeloid leukemia (AML)
Measurement of study drug concentrations to characterize pharmacokinetics. | 1 year
  - Determination of PK of elesclomol and elesclomol metabolites in subjects with relapsed or refractory acute myeloid leukemia (AML).

SECONDARY OUTCOMES:
Assessment of Dose Limiting Toxicities and Response based on Peripheral Blood Counts and Bone Marrow | 1 year
  - Determine the optimal Phase II dose and preliminary activity for elesclomol sodium in subjects with acute myeloid leukemia (AML).

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada